CLINICAL TRIAL: NCT02040805
Title: Comparison of Peer Facilitated Support Group and Cognitive Behavioral Therapy for Hoarding Disorder
Brief Title: Comparison of Treatment for Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE-1304-6000
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hoarding Disorder
Keywords: compulsive hoarding; clutter; hoarding disorder
MeSH Terms: conditions — Hoarding Disorder; Speech Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm parallel clinical trial with assessments pre- and post-treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Cognitive-Behavioral Therapy (Experimental): Sixteen sessions of group therapy facilitated by a psychologist.
  Interventions: Behavioral: Group Cognitive Behavioral Therapy
- Peer Facilitated Support Group (Experimental): Fifteen sessions of peer-facilitated group support.
  Interventions: Behavioral: Peer Facilitated Support Group

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — Group therapy over approximately 20 weeks, based on a structured manual adapted from the individual CBT workbook for hoarding by Steketee and Frost (2006). Each session will be 2 hours in length and consists of weekly check-ins, psychoeducation about hoarding, developing understanding and awareness of one's hoarding symptoms and patterns, behavior modification, cognitive restructuring, goal-setting, motivational enhancement, in vivo and imaginal exposure for discarding and acquisition, executive skills training (organization, sorting, planning, decision-making, problem-solving, etc.), guidelines on establishing "clutter buddies", and relapse prevention. Groups will be led by clinical postdoctoral psychology fellows in the Department of Psychiatry at UCSF.
  Arms: Group Cognitive-Behavioral Therapy
Behavioral: Peer Facilitated Support Group — Fifteen sessions of peer facilitated, group support, over the course of 20 weeks, based on a structured manualized approach (Buried in Treasures: Help for Compulsive Acquiring, Saving, and Hoarding). Each session will be 2 hours in length. In this model, two trained peers, usually, but not necessarily, with personal lived experience of hoarding, will guide the group chapter by chapter through the Buried in Treasures manual.
  Arms: Peer Facilitated Support Group

SUMMARY:
This study proposes to compare two forms of treatment for Hoarding Disorder (HD), a common and impairing neuropsychiatric syndrome that has a profound impact on the lives and functioning of individuals, families, and society. Specifically, we will compare a novel community-based group treatment led by individuals from the community who are not mental health professionals to the current standard of care treatment for Hoarding Disorder, Cognitive Behavioral Therapy, conducted by psychologists in a group setting. We hypothesized that both treatment types will be similarly effective in reducing hoarding severity.

DETAILED DESCRIPTION:
The study design for this proposal is a stratified, randomized, single-blind, non- inferiority trial comparing the current standard of care for treatment of Hoarding Disorder (HD), Group Cognitive Behavioral Therapy (G-CBT), to an innovative and promising community-based treatment, Group Buried in Treasures (G-BiT). Participants will be stratified by gender, psychiatric status (high vs. low burden of psychiatric symptoms) and insurance status (insured vs. under- or un-insured) so that equal numbers of individuals with each of these characteristics are randomized to each treatment arm. They will then be randomly assigned (randomized) to either G-CBT or G-BiT. Participants will know which treatment group they are assigned to, but those members of the research team who are conducting clinical or neuropsychological assessments or analyzing the data will not; they will be blinded to participant group assignment, and group leaders will be blinded to the psychiatric status, neurocognitive status, insurance status, etc, of participants. The study is a non-inferiority trial, that is, the hypothesis to be tested is that G-BiT is as effective, or no less effective, than G-CBT. We chose a non-inferiority design because we have no reason to believe G-BiT is better than G-CBT and our preliminary data, as well as outcomes previously reported for G- CBT and G-BiT, suggest that these treatments may have similar efficacies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hoarding Disorder

Exclusion Criteria:

* Individuals with active psychosis, schizophrenia, intellectual disability, or known dementia will be excluded
* Individuals who have participated in either cognitive-behavioral therapy for hoarding (group or individual) or in group Buried in Treasures in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Mathews, MD, Principal Investigator — University of Florida; Kevin L. Delucchi, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Mental Health Association, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred during April 2014 through February 2016. Participants were individuals with Hoarding Disorder recruited primarily through the Mental Health Association - San Francisco and flyers in the bay area (e.g. community center boards, coffee shops, laundry mats, libraries).
Period: Overall Study
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group
Started | 160 | 163
Completed | 118 | 113
Not Completed | 42 | 50
Not completed — Lost to Follow-up | 14 | 9
Not completed — Withdrawal by Subject | 28 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group | Total
Number analyzed (Participants) | 160 | 163 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.9) | 58.9 (10.6) | 59.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 124 | 241
  Male | 43 | 39 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 322 of the 323 randomized participants provided race/ethnicity information.
  Participants
    Race/Ethnicity Characteristics: number analyzed (Participants) | 160 | 162 | 322
    Race/Ethnicity Characteristics: American Indian/Alaskan Native | 0 | 1 | 1
    Race/Ethnicity Characteristics: Asian | 16 | 17 | 33
    Race/Ethnicity Characteristics: Black/African American | 17 | 6 | 23
    Race/Ethnicity Characteristics: Hispanic | 9 | 8 | 17
    Race/Ethnicity Characteristics: Native Hawaiian/Other Pacific Islander | 2 | 1 | 3
    Race/Ethnicity Characteristics: Other or Multiracial | 23 | 23 | 46
    Race/Ethnicity Characteristics: White | 89 | 101 | 190
    Race/Ethnicity Characteristics: Prefer not to answer | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Saving Inventory-Revised (SI-R)
Description: This is a 23-item self-report questionnaire that measures hoarding symptoms and their impact, including problems with acquisition, clutter, and difficulty discarding, as well as distress and impairment/interference. The SI-R is scored on a scale of 0-92. Higher scores indicate more severe hoarding, and scores of 42 and over are considered clinically significant hoarding. Although subscale scores can be calculated, this study uses total scores as the primary outcome.
Time Frame: Administered at screening before start of treatment groups and after last treatment group (20 weeks later).
Population: All randomized participants who were not lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group
Number analyzed (Participants) | 160 | 163
units on a scale
  Baseline | 64.5 (11.7) | 66.4 (11.6)
  End of Treatment: 20 weeks later: number analyzed (Participants) | 128 | 119
  End of Treatment: 20 weeks later | 45.9 (15.0) | 47.8 (14.2)
Statistical Analysis 1: Comparison: Group Cognitive-Behavioral Therapy vs Peer Facilitated Support Group; Test of non-inferiority; Test type: Non-Inferiority — Margin based on clinically meaningful change of >= 5 points; p = 0.04, t-test, 1 sided

2. Secondary Outcome: Activities of Daily Living Scale, Hoarding (ADL-H)
Description: The ADL-H is a 15-item self-report questionnaire that measures hoarding specific difficulties or problems that may impact daily functioning. It includes questions on activities affected by clutter or hoarding, problems in the home, and safety issues. For this study, the score on each ADL-H item was summed to create a total score ranging from 0 to 75. Higher scores indicate more severe functional impairment due to hoarding.
Time Frame: Administered at baseline and after last treatment group (20 weeks later).
Population: All randomized participants who were not lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group
Number analyzed (Participants) | 160 | 163
units on a scale
  Baseline: number analyzed (Participants) | 157 | 159
  Baseline | 29.9 (9.5) | 32.0 (11.2)
  End of Treatment: 20 weeks later: number analyzed (Participants) | 127 | 119
  End of Treatment: 20 weeks later | 25.5 (10.1) | 26.1 (8.7)
Statistical Analysis 1: Comparison: Group Cognitive-Behavioral Therapy vs Peer Facilitated Support Group; Test of non-inferiority; Test type: Non-Inferiority — Margin based on clinically meaningful change of >= 2.5 points; p = 0.05, t-test, 1 sided

3. Post Hoc Outcome: Longitudinal Follow-Up: Saving Inventory-Revised (SI-R)
Description: This is a 23-item self-report questionnaire that measures hoarding symptoms and their impact, including problems with acquisition, clutter, and difficulty discarding, as well as distress and impairment/interference. Using the SI-R, we obtained longitudinal follow-up data (defined as a second post-treatment assessment of hoarding symptom severity at least three months following completion of treatment). The total SI-R score was used, which ranges from 0-92, higher scores indicating more severe hoarding.
Time Frame: The post-hoc longitudinal data were collected at varying time points, but at least three months after the treatment ended. The range was 3 months to 25 months, with a mean of 14 months after treatment end.
Population: All randomized participants who were not lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group
Number analyzed (Participants) | 101 | 82
units on a scale | 48.2 (14.9) | 47.9 (13.9)
Statistical Analysis 1: Comparison: Group Cognitive-Behavioral Therapy vs Peer Facilitated Support Group; Test type: Other — linear mixed models analysis; p < 0.0001, Mixed Models Analysis; df=1

4. Post Hoc Outcome: Longitudinal Follow-Up: Activities of Daily Living Scale, Hoarding (ADL-H)
Description: The ADL-H is a 15-item self-report questionnaire that measures hoarding specific difficulties or problems that may impact daily functioning. It includes questions on activities affected by clutter or hoarding, problems in the home, and safety issues. Using the ADL-H, we obtained longitudinal follow-up data (defined as a second post-treatment assessment of hoarding specific difficulties or problems that may impact daily functioning at least three months following completion of treatment). For this study, a total score using the sum of all of the items was created, ranging from 0 to a total possible of 75. Higher scores indicate more severe impairment due to hoarding.
Time Frame: Post-hoc longitudinal analyses were conducted at three or more months' following the end of treatment. The range was 3-25 months, and the mean time to longitudinal follow up was 14 months.
Population: All randomized participants who were not lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group
Number analyzed (Participants) | 98 | 80
units on a scale | 27.6 (11.6) | 27.8 (9.7)
Statistical Analysis 1: Comparison: Group Cognitive-Behavioral Therapy vs Peer Facilitated Support Group; Test type: Other — linear mixed model; p < 0.0001, Mixed Models Analysis; df=1

ADVERSE EVENTS:
Arm/Group | Group Cognitive-Behavioral Therapy | Peer Facilitated Support Group
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/163
Other Adverse Events (participants affected / at risk) | 1/160 | 2/163
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group Cognitive-Behavioral Therapy (N=160) | Peer Facilitated Support Group (N=163)
Voluntary hospitalization due to "alcohol detox" "possible suicidality" (Psychiatric disorders) | 1 | 0 — Unanticipated hospitalization due events occurring in participant's life (event possibly related to study, but alternative cause is more likely)
Suicidality (Psychiatric disorders) | 0 | 1 — Participant became transiently suicidal while completing a homework assignment related to study.
Participant Fell (Social circumstances) | 0 | 1 — During a group session, a participant unintentionally walked into an obstruction and fell onto a chair.

LIMITATIONS AND CAVEATS:
The primary limitation in this study was loss to follow up. Additionally, the longitudinal follow-up assessment was post-hoc rather than being planned prior to study initiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No